CLINICAL TRIAL: NCT06820320
Title: Oral Iohexol in the Management of Chylous Ascites After Retroperitoneal or Extended Lymphadenectomy for Abdominal or Pelvic Malignant Tumor: an Innovative and Convenient Treatment
Brief Title: Oral Iohexol in the Management of Chylous Ascites After After Retroperitoneal or Extended Lymphadenectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No, 24/368-4648
Record Dates: First submitted 2025-01-16; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Chylous Ascites; Abdominal Neoplasm; Pelvic Neoplasms; Retroperitoneal Lymph Node Metastasis; Retroperitoneal Lymphadenectomy; Extended Lymphadenectomy
Keywords: Oral Iohexol; Chylous Ascites; Retroperitoneal Lymphadenectomy; Extended Lymphadenectomy; Abdominal Malignant Tumor; Pelvic Malignant Tumor
MeSH Terms: conditions — Chylous Ascites; Abdominal Neoplasms; Pelvic Neoplasms | interventions — Iohexol; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- oral iohexol group (Experimental)
  Interventions: Drug: oral iohexol; Procedure: Lymphangiography and Embolization

INTERVENTIONS:
Drug: oral iohexol — Upon diagnosing chylous ascites, patients received oral iohexol treatment, a critical intervention in our therapeutic armamentarium. The initial oral dose was standardized to ensure a balance between efficacy and patient safety. In the event of a less than optimal response or significant drainage within the first 24 hours, a second identical dose of Iohexol was considered to maintain therapeutic concentration levels in the body.
Procedure: Lymphangiography and Embolization — When conservative methods fall short in resolving chylous ascites, our protocol advances to precise interventional treatments. The escalation begins with ultrasound-guided lymphangiography. Through unilateral or bilateral inguinal lymph node access, iodized oil contrast is infused via a 9 ml/hour micro-pump, meticulously monitored by fluoroscopic imaging at 3-5 minutes intervals.
  Following precise localization of the leakage site, embolization is performed with a sequence of carefully calibrated steps. The process entails cone-beam CT scanning and 3D reconstruction for a clear depiction of the leak, followed by direct needle access to the lymphatic rupture under DSA guidance. A fine guidewire is inserted above the rupture, which facilitates the delivery of an embolizing mixture of iodized oil and NBCA glue. This is done with the utmost precision to prevent any spillage, ensuring the embolization's success and marking the conclusion of the procedure.

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of oral iohexol in the treatment of postoperative chylous ascites. It will also learn about the safety of oral iohexol. The main questions it aims to answer are:

* Confirm the potential of oral iohexol as an innovative therapeutic regimen.
* Confirm its ability to improve clinical outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 75 years;
* Patients underwent retroperitoneal or extended lymphadenectomy for abdominal or pelvic malignant tumors;
* Patients diagnosisted with postoperative Chylous ascites. Chylous ascites were defined by the presence of non-infectious, milky, or creamy effluent in drainage tubes surpassing 200 mL daily, paired with triglyceride concentrations exceeding 110 mg/dL

Exclusion Criteria:

* Patients with severe cardiac, hepatic and renal insufficiency;
* Patients with a history of iohexol allergy or allergy to contrast media;
* Patients who have received other interventions;
* Patients with severe intestinal obstruction or intestinal perforation;
* Patients who are unable to comply with the requirements of the study or are unable to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
grading system for efficacy of iohexol intervention | up to 3 weeks after the intervention
  The clinical responses post-Iohexol administration were evaluated against a set grading system:Grade A Success: This grade was assigned to patients who achieved complete cessation of lymphatic drainage with no clinical evidence of chylous ascites by the end of the first week post-treatment. To further ascertain the rapid action of Iohexol, 'Grade A+ Success' was defined for scenarios where this resolution occurred within the initial 3 days post-intervention. Grade B Success: Representing a substantial but partial therapeutic response, Grade B was denoted for patients who exhibited more than a 50% reduction in baseline lymphatic drainage within the first week, but did not meet the criteria for Grade A success. Non-responders: Patients who did not conform to the criteria for Grade A or B success were categorized as non-responders. This group was identified for further evaluation and considered for additional treatment modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grist TM, Canon CL, Fishman EK, Kohi MP, Mossa-Basha M. Short-, Mid-, and Long-term Strategies to Manage the Shortage of Iohexol. Radiology. 2022 Aug;304(2):289-293. doi: 10.1148/radiol.221183. Epub 2022 May 19. PMID 35587228